CLINICAL TRIAL: NCT03196804
Title: A Dose Blocked-randomized, Double-blind, Placebo-controlled, Multiple Dosing and Dose-escalation Phase I Clinical Trial to Investigate the Safety, Tolerability and Pharmacokinetic Characteristics of LC28-0126 in Healthy Male Subjects
Brief Title: A Phase I Clinical Trial to Investigate the Safety, Tolerability and Pharmacokinetic Characteristics of LC28-0126.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LG Chem (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LG-CYCL003
Record Dates: First submitted 2017-06-20; First posted 2017-06-23 (Actual); Last update posted 2018-04-11 (Actual); Status verified 2018-04

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LC28-0126 (Experimental): LC28-0126(IV)
  Interventions: Drug: LC28-0126
- Placebo (Placebo Comparator): Placebo of LC28-0126
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LC28-0126 — LC28-0126
  Arms: LC28-0126
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
To assess the safety, tolerability and pharmacokinetic characteristics of LC-28-0126 multiple iv injection in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects between the ages of 19 and 45 years at screening.
* Subjects with BMI between 18.0(inclusive) and 27.0 kg/m2 (exclusive); and a total body weight between 55 kg (inclusive) and 90 kg (exclusive)

Exclusion Criteria:

* Participation in a clinical research study within the previous 3 months
* Regular alcohol consumption >21 units per week.

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2017-06-07 (Actual); Primary Completion 2017-11-15 (Actual); Study Completion 2017-11-15 (Actual)

PRIMARY OUTCOMES:
Adverse events | 18 days

SECONDARY OUTCOMES:
Cmax | up to 6 days post-dose
AUC | up to 6 days post-dose

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Clinical Trial Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim E, Hwang I, Lee S, Oh J, Chung H, Jin M, Kim SH, Yu KS. Pharmacokinetics and Tolerability of LC28-0126, a Novel Necrosis Inhibitor, After Multiple Ascending Doses: A Phase I Randomized, Double-blind, Placebo-controlled Study in Healthy Male Subjects. Clin Ther. 2020 Oct;42(10):1946-1954.e2. doi: 10.1016/j.clinthera.2020.08.011. Epub 2020 Sep 24. PMID 32980184